CLINICAL TRIAL: NCT03234530
Title: Linking the Effects of 9/11 to Kidney Disease
Brief Title: World Trade Center Kidney-Link
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Maryann Mclaughlin, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 16-0899; U01OH011326-01A1 (NIH)
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Chronic Kidney Diseases; Obstructive Sleep Apnea
Keywords: albuminuria; sleep apnea; particulate matter; renal injury
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sleep Apnea, Obstructive; Albuminuria; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, plasma, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WTC responders: WTC Health Program participants
- Urban workers: Control group of urban workers in NYC not exposed to the dust from the WTC

SUMMARY:
This study focuses on the prevalence and identification of kidney disease among participants of the WTC Health Program and the study team are planning to assess kidney disease in a multi-factorial manner. The first aim of this study is to correlate kidney dysfunction with 9/11 exposure, and the study team predicts that exposure to 9/11 is an independent risk factor in kidney disease among the WTC Health Program participants. Secondly, the study team proposes that a well-established WTC-related condition, obstructive sleep apnea (OSA), is independently associated with kidney disease. In addition, the study team believe there is a temporal causative relationship between evidence of kidney disease and the severity of OSA. Finally, the last aim is to further identify and explore potential mechanisms and phenotypes of kidney disease in participants of the WTC Health Programs.

Regardless of whether the analyses support or reject these hypotheses, the findings will be of equally great public health importance. Successful completion of the proposed research would address a critical knowledge gap regarding the risk of kidney damage among this group of patients, and would inform future mechanistic studies with the potential to impact prevention.

DETAILED DESCRIPTION:
Exposure to environmental toxins results in significant long-term health effects in workers. More than 91,000 rescue and recovery workers and volunteers at the World Trade Center (WTC) sustained exposure to thousands of tons of coarse and fine particulate matter. Thousands of responders are currently treated for WTC-related health conditions or may be at risk for worsening health. Toxic effects of particulate matter are known to affect the pulmonary, renal and cardiovascular systems. The specific effects of the exposure to 9/11 are partly known, and require further investigation, as outlined in the Zadroga Act (Public Law111-347).

This study builds on the preliminary data to address a critical knowledge gap about the risk of kidney damage among WTC responders, the progression of kidney decline since exposure, and the association of kidney disease with a defined WTC-related diagnosis, obstructive sleep apnea (OSA). Successful completion of the proposed research would address a critical knowledge gap regarding the risk of kidney damage and the relationship to important chronic diseases (OSA and immune-mediated disease) among WTC participants, and would inform future mechanistic studies with the potential to impact disease prevention.

Specific Aim 1: To quantify the risk of kidney damage and the relationship to 9/11 exposure among WTC Health Program participants. Currently, the cohort of 406 first responders represents the sole dedicated evaluation of kidney disease in WTC Health Program participants. The study team will test the hypothesis that exposure to 9/11 is independently associated with kidney disease and enrich the enrollment of the current study population with a diversified population including categories of workers who have not been enrolled, as well as a control group of urban workers (NYC) not exposed to the dust from the WTC.

Aim 1a. The study team hypothesize that albuminuria and decreased estimated glomerular filtration rate (eGFR) will occur more frequently in WTC responders than in the general population and will correlate with the degree of exposure as defined by the previously defined WTC exposure score (adjusting for demographics, family history of chronic kidney disease (CKD), and diagnosed, treated or laboratory confirmed diabetes and hypertension). The study team will also assess established urine biomarkers of proximal tubular injury, including β2-M, Kidney Injury Molecule-1 (KIM-1), and Interleukin 18 (IL-18), as well as markers of distal tubular function, Loop of Henle function, and tubulointerstitial inflammation.

Aim 1b. The study team hypothesize that initial exposure to 9/11 contributed to reduction in renal function over time. The study team will quantify change in renal function over time by analyzing eGFR at WTC Health Program Visit 1 (V1) and subsequent visits, adjusting for known co-morbid conditions.

Aim 1c. The study team will create a repository of WTC responders with established kidney disease (including relatively rare disease) to qualitatively evaluate and describe the spectrum of kidney disease in the entire WTC population and compare to patterns of kidney disease in the general population. The study team will actively enlist those with a verified physician diagnosis of kidney disease, and collect biopsy reports and slides for review.

Specific Aim 2: Evaluate the association of kidney disease and the established WTC-related condition, OSA.

Aim 2a. OSA is particularly prevalent among WTC cohorts. The study team hypothesize that there is an independent association between prevalent OSA and prevalent kidney disease.

Aim2b. The study team hypothesize that OSA independently contributes to the progression of kidney disease. The study team will assess the temporal relationship of eGFR decline to the presence and severity of OSA, using longitudinal data from the WTC data center.

Specific Aim 3: To evaluate potential mechanisms of kidney injury in WTC Health Program participants.

Aim3a. In order to understand the role of chronic inflammation, the study team will evaluate established inflammatory markers which have been implicated as potential mediators of both OSA and CKD, including IL-10, IL-13, IL-1β, IL-2, IL-4, IL-6, IL-8, TNF-α, IFN-γ, IL-12p70., high sensitivity C-reactive protein (hs-CRP), and white blood cell count (WBC).

Aim3b. Based on the preliminary data noting increases in heavy metal levels in urine and blood, the study team will narrow the focus to evaluate the role of cadmium and lead in the development of kidney disease with evaluations of lead content in bone (marker of long-term exposure) as well as in blood. Since study participants include law enforcement personnel (with known exposure to lead), the characterization of bone lead levels will have an important health impact, whether or not a relationship to 9/11 is detected.

Aim3c. In a registry cohort of WTC responders with established kidney disease the study team will explore potential mechanisms as determined by the observed patterns of disease by developing a comprehensive repository of data on WTC Health Program participants with common and rare kidney diseases, the study team will define specific clinical profiles and identify potential mechanisms that warrant future study. Importantly, the study team will develop a process across all WTC Health Programs (inclusive of approximately 50,000 individuals), to monitor those with early kidney disease as well as those with biopsy-proven kidney disease, at any stage.

ELIGIBILITY:
Inclusion Criteria:

- Exposed Group: - Adult patients (35 to 75 years)

* Enrolled or was seen at any of the WTC Clinical Centers of Excellence

Unexposed Group: - Adult patients (35 to 75 years)

* Lived or worked in NYC at least 10 years since 9/11/01 but were not exposed to the the dust at Ground Zero (not living in proximity of Ground Zero, nor involved in the rescue and recovery at Ground Zero

Registry Part: - Adult patient (18 to 75 years)

* Enrolled or was seen at any of the WTC Clinical Centers of Excellence or WTC Environmental Health Centers
* With a diagnosis of any Kidney Injury or disease after 9/11/01

Exclusion Criteria:

* Patients below 18 years of age
* Individuals with an occupation involving chronic exposure to inhaled particulate matter (e.g. iron/steel workers and sand hog workers)
* For the registry part, patients with kidney disease prior to 9/11/01

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: World Trade Center rescue and recovery workers and volunteers who are enrolled or being seen in any WTC Clinical Centers of Excellence
Sampling Method: Non-Probability Sample
Enrollment: 555 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
glomerular filtration rate (eGFR) | day 1
  eGFR will be calculated using the Chronic Kidney Disease Epidemiology Consortium (CKD-EPI) equations. The proposed studies will evaluate differences in the combined creatinine-cystatin C eGFR, which provides the most accurate estimate of GFR, and the creatinine-based CKD-EPI eGFR, which is more practical for use in clinical practice and in monitoring programs. Values > 200 will be set to 200mL/min/1.73m2
albuminuria | day 1
  albumin level in urine

SECONDARY OUTCOMES:
Berlin questionnaire | day 1
  Those who are not diagnosed with sleep apnea will be assessed for risk of developing sleep apnea using the Berlin questionnaire. It includes 11 questions organized into three categories, 5 questions related to snoring and the cessation of breathing in category 1, 4 questions related to daytime sleepiness in category 2, 1 question about high blood pressure, and 1 question regarding BMI in category 3. When two of three categories are classified as positive for a patient, the patient is rated as being at high risk of having OSA.
apnea-hypopnea index (AHI) | day 1
  Those at high risk for sleep apnea will undergo home sleep a study test to determine apnea hypopnea index (AHI).
  Those diagnosed with sleep apnea, latest sleep study will be used to obtain AHI. To determine AHI, add the total number of apnea events, plus hypopnea events and divide by the total number of minutes of actual sleep time, then multiply by 60. AHI - Apnea Hypopnea Index - The # of apneas and hypopneas per hour.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann McLaughlin, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The final research data will be a computerized dataset and includes self-reported demographic and medical data, responses from standard questionnaires, as well as results of laboratory tests (urine and blood samples) . Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.